CLINICAL TRIAL: NCT05949164
Title: The IPAd Study: Exploring the Association Between Insomnia and Positive Airway Pressure Adherence in Children
Acronym: IPAd
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Indra Narang, Professor, The Hospital for Sick Children
Other Study IDs: 1000080572
Record Dates: First submitted 2023-06-24; First posted 2023-07-17 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea; Hypoventilation; Central Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypoventilation; Sleep Apnea, Central | interventions — Prion Proteins

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Children able to answer questionnaires independently: Children who are deemed by a healthcare professional to be able to answer questionnaires independently (group 1) will be asked to complete self-reported questionnaires. Caregivers will also be asked to complete proxy-reported questionnaires.
  Interventions: Behavioral: Insomnia
- Group 2: Children unable to answer questionnaires: The caregivers of children who are deemed by a healthcare professional to be unable to answer questionnaires (group 2) will be invited to complete proxy-reported questionnaires only. There are no self-reported questionnaires for this group.
  Interventions: Behavioral: Insomnia

INTERVENTIONS:
Behavioral: Insomnia — The primary exposure is insomnia

SUMMARY:
Sleep-disordered breathing (SDB) is prevalent in children and adolescents and untreated SDB impacts key indicators of physical and psychosocial health. Positive airway pressure (PAP) therapy is highly effective for the treatment of SDB and is associated with favorable clinical outcomes but is limited by poor adherence. Emerging literature in adults suggests that intolerance to PAP therapy may be related to coexisting insomnia. However, the presence of insomnia in children with known SDB as well as its impact on PAP adherence have not been explored. This proposal will explore the association of coexisting insomnia on PAP adherence in children with SDB using a cross-sectional study design. The investigators will assess the association between insomnia and PAP therapy adherence, measured as the mean minutes of nightly PAP usage over 6 months of use on objective downloads.

DETAILED DESCRIPTION:
Sleep-disordered breathing (SDB) is prevalent in children and adolescents and untreated SDB impacts key indicators of physical and psychosocial health. Positive airway pressure (PAP) therapy is highly effective for the treatment of SDB and is associated with favorable clinical outcomes but is limited by poor adherence. Emerging literature in adults suggests that intolerance to PAP therapy may be related to coexisting insomnia. This study addresses a critical knowledge gap regarding the association between insomnia and PAP therapy adherence amongst children with SDB. These results will inform future prospective studies on targeted effective interventions to improve PAP adherence in children with SDB.

SDB encompasses a range of breathing disorders during sleep including obstructive sleep apnea (OSA), central sleep apnea (CSA), and hypoventilation. PAP therapy is a common treatment modality for SDB that is often implemented after targeted treatment strategies do not fully cure SDB. PAP therapy, which delivers pressurised air via nasal or oronasal interfaces, effectively distends the upper airway to ameliorate OSA and can assist ventilation with pressure support breaths. PAP is highly efficacious when used on a nightly basis and is typically required for many years into adulthood. The use of PAP has been associated with increased survival and improved health-related quality of life in people with neuromuscular disease. However, SDB remains undertreated or untreated in many children due to poor adherence. A deeper understanding of associations with PAP adherence across the diagnostic spectrum may yield greater benefits for all children on PAP therapy.

Insomnia is highly prevalent in childhood, occurring in up to 37% of children. Insomnia is associated with reduced cognition and academic functioning as well as reduced health-related quality of life, substance use, and increased risk of psychiatric problems. There is emerging evidence that insomnia commonly coexists with OSA in children. A bi-directional causal relationship likely exists whereby OSA is exacerbated by sleep fragmentation, hyper-arousal, and modified sleep architecture associated with insomnia whereas insomnia symptoms are induced by repeated post-obstruction awakenings in OSA. Of importance is that coexisting insomnia and OSA is associated with greater morbidity than either condition alone. To date, there is minimal reported literature on coexisting insomnia with other SDB including CSA and nocturnal hypoventilation. Although similar pathophysiological mechanisms may exist for CSA, there has been little reported in the literature regarding these relationships.

More recently, insomnia has been identified as a risk factor for reduced PAP therapy adherence rates in adult populations due to hypersensitivity to PAP equipment side effects, early discontinuation of therapy, and reduced sleep duration. The impact of insomnia on PAP adherence has never been explored in children. Further, the impact of insomnia on PAP adherence in populations with other SDB diagnoses other than OSA has yet to be explored. Elucidating the impact of coexisting insomnia on PAP adherence may inform future targeted management strategies to improve PAP adherence, such as the addition of cognitive behavioral therapy, and may lead to improved outcomes in children with SDB.

ELIGIBILITY:
Participant Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Children aged 4-17 years old
2. Prescribed PAP therapy for at least 6 months

Participant Exclusion Criteria

An individual or caregiver who meets one or more of the following criteria will be excluded from participation in this study:

1) Limited knowledge and proficiency in English to complete the study as judged by the clinical team.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents established on PAP therapy
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
PAP therapy adherence | 6 months
  PAP therapy adherence measured as the mean minutes of nightly PAP usage over 6 months

SECONDARY OUTCOMES:
PAP therapy adherence | 6 months
  PAP therapy adherence expressed as a percentage of total sleep time
PAP therapy adherence | 3 months
  PAP therapy adherence measured as the mean minutes of nightly PAP usage over 3 months
PAP therapy adherence | 3 months
  PAP therapy adherence expressed as a percentage of total sleep time
PAP therapy adherence | 2 weeks
  PAP therapy adherence measured as the mean minutes of nightly PAP usage over 2 weeks
PAP therapy adherence | 2 weeks
  PAP therapy adherence expressed as a percentage of total sleep time
PAP therapy adherence | 3 months
  PAP therapy adherence expressed as a dichotomous outcome (PAP usage for at least 4 hours per night for 70% of nights)
PAP therapy adherence | 3 months
  PAP therapy adherence expressed as a dichotomous outcome (PAP usage for at least 6 hours per night for 70% of nights)
PAP therapy adherence | 6 months
  PAP therapy adherence expressed as a dichotomous outcome (PAP usage for at least 4 hours per night for 70% of nights)
PAP therapy adherence | 6 months
  PAP therapy adherence expressed as a dichotomous outcome (PAP usage for at least 6 hours per night for 70% of nights)
Physical Well-being (percentage rank) | 1 week
  The Physical Well-being Scale from the KIDSCREEN-27 questionnaire will be used. The percentage rank range is 0-100, with lower scores indicating lower physical well-being.
Psychological Well-being (percentage rank) | 1 week
  The Psychological Well-being Scale from the KIDSCREEN-27 questionnaire will be used. The percentage rank range is 0-100, with lower scores indicating a "dissatisfaction with life".
Autonomy and Parent Relation (percentage rank) | 1 week
  The Autonomy and Parent Relation Well-being Scale from the KIDSCREEN-27 questionnaire will be used. The percentage rank range is 0-100, with lower scores indicating lower autonomy.
Self-Perception (percentage rank) | 1 week
  The Self-Perception Scale from the KIDSCREEN-27 questionnaire will be used. The percentage rank range is 0-100, with lower scores indicating lower self-perception.
Social Support and Peers (percentage rank) | 1 week
  The Social Support and Peers Scale from the KIDSCREEN-27 questionnaire will be used. The percentage rank range is 0-100, with lower scores indicating lower social support.
Daytime Sleepiness | 1 month
  The Epworth Sleepiness Scale is scored from 0-24, with higher scores indicating greater sleepiness.
Depressive Symptoms (T-score) | 7 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Item Bank v2.0 - Depressive Symptoms Questionnaire generates a T-score. Higher scores indicate increased depressive symptoms (patient-reported questionnaire range 35.2-82.4).
Depressive Symptoms (T-score) | 7 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy Bank v2.0 - Depressive Symptoms Questionnaire generates a T-score. Higher scores indicate increased depressive symptoms (proxy-reported questionnaire range 36.2-84.7).
Anxiety Symptoms (T-score) | 7 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Bank v2.0 - Anxiety Questionnaire generates a T-score. Higher scores indicate increased anxiety symptoms (patient-reported questionnaire range 33.5-83.3).
Anxiety Symptoms (T-score) | 7 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy Bank v2.0 - Anxiety Questionnaire generates a T-score. Higher scores indicate increased anxiety symptoms (proxy-reported questionnaire range 34.6-86.4).
Chronotype | 4 week
  Measured with the Children's Chronotype Questionnaire. The chronotype categorizations including morningness, eveningness, and neither.
Chronotype | 4 week
  Measured with the Reduced Morningness-Eveningness questionnaire. The chronotype categorizations including morningness, eveningness, and neither.
Chronotype | 4 week
  Measured with the Munich Chronotype Questionnaire for Children and Adolescents. The chronotype categorizations including morningness, eveningness, and neither.
Mid-Sleep Point | 4 week
  Measured with the Munich Chronotype Questionnaire for Children and Adolescents
Mid-Sleep Point | 4 week
  Measured with the Children's Chronotype Questionnaire
Sleep Hygiene (total score) | 1 month
  The Adolescent Sleep Hygiene Scale total score ranges from 1-6. Higher scores indicate better success with sleep hygiene.
Sleep Hygiene (Physiological Factor) | 1 month
  Subscale from the Adolescent Sleep Hygiene Scale total score. The score ranges from 1-6. Higher scores indicate better success with sleep hygiene.
Sleep Hygiene (Behavioral Arousal Factor) | 1 month
  Subscale from the Adolescent Sleep Hygiene Scale total score. The score ranges from 1-6. Higher scores indicate better success with sleep hygiene.
Sleep Hygiene (Cognitive/Emotional Factor) | 1 month
  Subscale from the Adolescent Sleep Hygiene Scale total score. The score ranges from 1-6. Higher scores indicate better success with sleep hygiene.
Sleep Hygiene (Sleep Environment Factor) | 1 month
  Subscale from the Adolescent Sleep Hygiene Scale total score. The score ranges from 1-6. Higher scores indicate better success with sleep hygiene.
Sleep Hygiene (Sleep Stability Factor) | 1 month
  Subscale from the Adolescent Sleep Hygiene Scale total score. The score ranges from 1-6. Higher scores indicate better success with sleep hygiene.
Sleep Hygiene (Daytime Sleep Factor) | 1 month
  Subscale from the Adolescent Sleep Hygiene Scale total score. The score ranges from 1-6. Higher scores indicate better success with sleep hygiene.
Sleep Hygiene (Substances Factor) | 1 month
  Subscale from the Adolescent Sleep Hygiene Scale total score. The score ranges from 1-6. Higher scores indicate better success with sleep hygiene.
Sleep Hygiene (Bedtime Routine Factor) | 1 month
  Subscale from the Adolescent Sleep Hygiene Scale total score. The score ranges from 1-6. Higher scores indicate better success with sleep hygiene.
Adherence Barriers to CPAP | 2 weeks
  The score range for the Adherence Barriers to CPAP Questionnaire is 31-155. Higher scores indicate more barriers.
Total Difficulties Score | 6 months
  The Strengths and Difficulties Questionnaire generates a total difficulties score ranging from 0-40, with higher scores indicating greater behavioral difficulty.
Emotional Problems Score | 6 months
  The Strengths and Difficulties Questionnaire generates an emotional problems score ranging from 0-10, with higher scores indicating greater difficulty.
Conduct Problems Score | 6 months
  The Strengths and Difficulties Questionnaire generates a conduct problems score ranging from 0-10, with higher scores indicating greater difficulty.
Hyperactivity Score | 6 months
  The Strengths and Difficulties Questionnaire generates a hyperactivity score ranging from 0-10, with higher scores indicating greater difficulty.
Peer Problems Score | 6 months
  The Strengths and Difficulties Questionnaire generates a peer problems score ranging from 0-10, with higher scores indicating greater difficulty.
Prosocial Score | 6 months
  The Strengths and Difficulties Questionnaire generates a prosocial score ranging from 0-10, with higher scores indicating greater prosocial behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Indra Narang, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No